CLINICAL TRIAL: NCT01028131
Title: A Computer-Assisted Brief Motivational Intervention for Smoking During Pregnancy: The Healthy Pregnancy Project (HPP)
Brief Title: Computer-Assisted Intervention for Smoking During Pregnancy
Acronym: HPP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Steven J. Ondersma, Associate Professor, Wayne State University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: R21DA021668-01 (NIH); R21DA021668-02 (NIH)
Record Dates: First submitted 2009-12-08; First posted 2009-12-09 (Estimated); Results first posted 2013-06-10 (Estimated); Last update posted 2013-06-10 (Estimated); Status verified 2013-06

CONDITIONS: Smoking
Keywords: cigarette smoking; pregnancy; intervention; efficacy; Motivational Interviewing; Contingency Management
MeSH Terms: conditions — Smoking; Cigarette Smoking | interventions — Crisis Intervention

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control (No Intervention): Participants randomized by the computer into this condition will only view the 20-minute video clips of music and tv videos.
- Computerized brief intervention (5As) (Experimental): After completing the brief assessment battery, participants will interact with the computer for approximately 20 minutes, with structure being based on the Five A model (ask, advise, assess, assist & arrange) and Motivational Interviewing.
  Interventions: Behavioral: Computer-delivered brief intervention (5As)
- Contingency Management Alone (Experimental): Participants randomized by the computer into this condition will view a 20-minute music and tv video clip after completing the brief assessment. The research assistant will then briefly describe the CM process, with some time to discuss questions regarding procedure to assure understanding. The CM condition will involve participant-initiated submission of urine samples at prenatal visits. Clinic staff will have no responsibility for the CM component other than calling research staff when a participant wishes to submit a sample. Clinic staff will not schedule any new, additional, or unnecessary prenatal visits.
  Interventions: Behavioral: Contingency Management
- Combined Brief Intervention and CM (Experimental): Combined intervention. Participants in this condition will receive both the brief intervention and the brief description of the CM process.
  Interventions: Behavioral: Computer-delivered brief intervention (5As); Behavioral: Contingency Management

INTERVENTIONS:
Behavioral: Computer-delivered brief intervention (5As) — After completing the brief assessment battery, participants will interact with the computer for approximately 20 minutes, with structure being based on the Five A model and Motivational Interviewing.
  Other Names: Brief intervention; 5As; Brief motivational intervention
  Arms: Combined Brief Intervention and CM; Computerized brief intervention (5As)
Behavioral: Contingency Management — Participants randomized by the computer into this condition will view a 20-minute music and tv videos after completing the brief assessment. The research assistant will then briefly describe the CM process, with a period for questions to assure understanding. The CM condition will involve participant-initiated submission of urine samples at prenatal visits. Clinic staff will have no responsibility for the CM component other than calling research staff when a participant wishes to submit a sample. Clinic staff will not schedule any new, additional, or unnecessary prenatal visits.
  Other Names: Voucher-based reinforcement
  Arms: Combined Brief Intervention and CM; Contingency Management Alone

SUMMARY:
This study will develop:

1. Develop the computer-based brief intervention and Contingency Management (CM) components, with repeated feedback from experts, prenatal clinic staff, and participants.
2. Recruit 110 pregnant women who are actively smoking, and randomly assign recruited women to Brief Intervention, CM, combined, or control conditions.
3. Conduct follow-up evaluation at 12 weeks post-intervention to measure self-reported smoking, breath carbon monoxide (CO), and urinary cotinine levels.
4. Collect data regarding birth outcomes and evaluate the feasibility of various methods of post-partum follow-up.

DETAILED DESCRIPTION:
Participants & Procedure

Women will be approached while in the waiting room of various clinics at the Detroit Medical Center. Clinic staff will inform patients of the study and its goals via a flyer that will be distributed at the reception window as women arrive for their appointments. If the women are interested, they will answer some questions and provide their contact information on the back of the flyer. Then they will place the flyer in a ballot box that is locked and only can be accessed by the Research Staff. Research staff may also be at the clinic to recruit women from the waiting room. When the research staff meets with potential participants. The study will be briefly described, and those indicating tentative interest will be screened for age and language ability (informally). Those indicating tentative interest, reporting age of at least 18 years, gestation 27 weeks or less, and demonstrating adequate ability to speak and understand spoken English will be brought to a nearby private room.

First, informed consent for screening will be obtained using an information sheet; this sheet will describe the purpose of the screening, and will emphasize that participation in the initial screening is anonymous. Those who agree will be given a very brief demonstration of the use of the computer, after which they will complete the brief (10-item) screener. All interactions with the computer will involve a touch-screen and headphones for private presentation of all information aurally as well as visually; in many previous studies, including pilot testing at this clinic, the software has been proven extremely easy to use, even for women lacking any prior computer experience. Those who endorse smoking cigarettes (even a puff) in the past week will be told of the full study in detail, and written informed consent will be sought (with a brief quiz to assure understanding). Those who provide consent will again interact directly with the computer.

Intervention

The computer itself will perform randomization and will gather all research data except for baseline breath CO (which is higher among persons who smoke), which will be obtained (via a Micro Smokerlyzer® from Bedfont Scientific Ltd.) and entered into the computer by the research staff. The entire process, including consent, will take approximately 40 minutes regardless of experimental condition (to which the research staff will be blind). Research staff will tell clinic staff of the patient's whereabouts so that the patient is not passed over when staff call her to an exam room; unfinished study procedures will be completed in the exam room prior to the physician's entrance, and/or after the appointment is completed.

Women (N = 110) who report smoking cigarettes (even a puff) during pregnancy will be randomly assigned to computer-based brief intervention alone, CM alone, brief intervention plus CM, or attention control conditions. Women randomly assigned to the computer-based intervention condition will receive an approximately 20-minute intervention modeled after motivational interviewing (MI).

Women randomly assigned to the CM condition will be told that, if they choose, they can ask to be tested (via provision of a urine sample) for smoking, up to five times, at a regularly scheduled prenatal visit. Research staff will conduct these tests.

8-Week Follow-Up

Women who enroll in the study will be contacted via mail and telephone, as necessary, to schedule a 8-week follow-up at the PI's lab or at the prenatal clinic, depending upon the participant's preference. Research staff completing follow-up testing will be kept blind to intervention condition. The primary outcome measure will be urinary cotinine-verified abstinence at follow-up; birth outcome data will also be gathered from hospital records. At follow-up, participants will (a) complete all measures on the computer again, (b) provide breath CO; (c) provide a final urine sample for testing of urinary cotinine (evidence of smoking).

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years
* pregnant, gestation <= 27 weeks
* cigarette smoking in the past week (even if only one puff)

Exclusion Criteria:

* inability to speak or understand spoken English
* do not intend to carry pregnancy to full term
* frank psychosis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2007-06; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Ondersma, PhD, Principal Investigator — Wayne State University
Locations (1):
- Wayne State University-Detroit Medical Center, Detroit, Michigan, United States

REFERENCES:
- [Derived] Ondersma SJ, Svikis DS, Lam PK, Connors-Burge VS, Ledgerwood DM, Hopper JA. A randomized trial of computer-delivered brief intervention and low-intensity contingency management for smoking during pregnancy. Nicotine Tob Res. 2012 Mar;14(3):351-60. doi: 10.1093/ntr/ntr221. Epub 2011 Dec 9. PMID 22157229

RESULTS

PARTICIPANT FLOW:
Groups:
- Computerized Brief Intervention (5As): After completing the brief assessment battery, participants will interact with the computer for approximately 20 minutes, with structure being based on the Five A model and Motivational Interviewing.
- Contingency Management Alone: Participants randomized by the computer into this condition will view a 20-minute music and tv video clip after completing the brief assessment. The research assistant will then briefly describe the CM process, with some time to discuss questions regarding procedure to assure understanding. The CM condition will involve participant-initiated submission of urine samples(looking for clean samples with cotinine less than 100 ng/ml) at prenatal visits. Clinic staff will have no responsibility for the CM component other than calling research staff when a participant wishes to submit a sample. Clinic staff will not schedule any new, additional, or unnecessary prenatal visits.
Period: Overall Study
Arm/Group | Control | Computerized Brief Intervention (5As) | Contingency Management Alone | Combined Brief Intervention and CM
Started | 26 | 26 | 28 | 30
Completed Intervention/Control Session | 26 | 26 | 28 | 30
Completed | 23 | 23 | 22 | 26
Not Completed | 3 | 3 | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Contingency Management Alone: Participants randomized by the computer into this condition will view a 20-minute music and tv video clip after completing the brief assessment. The research assistant will then briefly describe the CM process, with some time to discuss questions regarding procedure to assure understanding. The CM condition will involve participant-initiated submission of urine samples at prenatal visits (looking for clean samples - cotinine less than 100 ng/ml). Clinic staff will have no responsibility for the CM component other than calling research staff when a participant wishes to submit a sample. Clinic staff will not schedule any new, additional, or unnecessary prenatal visits.
- Total: Total of all reporting groups
Arm/Group | Control | Computerized Brief Intervention (5As) | Contingency Management Alone | Combined Brief Intervention and CM | Total
Number analyzed (Participants) | 26 | 26 | 28 | 30 | 110
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 26 | 26 | 28 | 30 | 110
  >=65 years | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 28.5 (7.5) | 25.8 (4.8) | 29.3 (6.7) | 27.7 (6.1) | 27.9 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 26 | 28 | 30 | 110
  Male | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 26 | 26 | 28 | 30 | 110

OUTCOME MEASURES:

1. Primary Outcome: Smoking Behavior (Self-report Confirmed by Expired Breath CO)
Description: All participants were analyzed as assigned. Total N was determined primarily by resource availability in this Stage Ib trial. Number represents number of abstinent participants in each condition.
Time Frame: 8 week follow up
Measure: Number; unit: participants
Groups:
- Contingency Management Alone: Participants randomized by the computer into this condition will view a 20-minute music and tv video clip after completing the brief assessment. The research assistant will then briefly describe the CM process, with some time to discuss questions regarding procedure to assure understanding. The CM condition will involve participant-initiated submission of urine samples at prenatal visits (looking for clean samples -cotinine less than 100 ng/ml). Clinic staff will have no responsibility for the CM component other than calling research staff when a participant wishes to submit a sample. Clinic staff will not schedule any new, additional, or unnecessary prenatal visits.
Arm/Group | Control | Computerized Brief Intervention (5As) | Contingency Management Alone | Combined Brief Intervention and CM
Number analyzed (Participants) | 23 | 23 | 22 | 26
participants | 2 | 7 | 2 | 5

2. Primary Outcome: Urinary Cotinine
Description: Cotinine, as measured by urine sample taken and follow-up. Measured as number of participants abstinent by cotinine analysis.
Time Frame: 8 week follow-up
Measure: Number; unit: participants
Arm/Group | Control | Computerized Brief Intervention (5As) | Contingency Management Alone | Combined Brief Intervention and CM
Number analyzed (Participants) | 23 | 23 | 22 | 26
participants | 4 | 10 | 3 | 4

ADVERSE EVENTS:
Groups:
- Contingency Management Alone: Participants randomized by the computer into this condition will view a 20-minute music and tv video clip after completing the brief assessment. The research assistant will then briefly describe the CM process, with some time to discuss questions regarding procedure to assure understanding. The CM condition will involve participant-initiated submission of urine samples at prenatal visits. Clean samples (cotinine less than 100 ng/ml) will result in the immediate provision of a $50 Target gift card. Clinic staff will have no responsibility for the CM component other than calling research staff when a participant wishes to submit a sample. Clinic staff will not schedule any new, additional, or unnecessary prenatal visits.
Arm/Group | Control | Computerized Brief Intervention (5As) | Contingency Management Alone | Combined Brief Intervention and CM
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26 | 0/28 | 0/30
Other Adverse Events (participants affected / at risk) | 0/26 | 0/26 | 0/28 | 0/30

LIMITATIONS AND CAVEATS:
Although all effects favored brief computer session, the small sample size limited our ability to detect small effects. The sample was almost exclusively low-income African-American women. Follow-up period was also, of necessity, relatively brief.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No